CLINICAL TRIAL: NCT02974452
Title: Age-related Changes in Activation Patterns of Shoulder Muscles
Brief Title: Age-related Changes of Shoulder Muscles
Acronym: SEMG
Status: Completed | Type: Observational
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Cristina Lirio Romero, Physiotherapist, University of Alcala
Other Study IDs: UAlcalaH
Record Dates: First submitted 2016-11-20; First posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Electromyography

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group I: Older adults: healthy subjects older than 68 years old whose shoulder muscle are measured by surface electromyography
- Group II: Adults: healthy subjects 43 to 67 years old, whose shoulder muscle are measured by surface electromyography
- Group III: Young adults: healthy subjects 20 to 42 years old, whose shoulder muscle are measured by surface electromyography

SUMMARY:
A cross-sectional descriptive study, in which the surface electromyographic activity of five shoulder muscles was compared in three populations: older adults, middle-aged adults and young adults. The evaluation of the electromyographic data offers a suitable foundation to understand aging process.

This supports that surface electromyography provide information about the aged shoulder muscles. Loss of functionality is suffered by a high percentage of older adults, which greatly limits their physical activity. In this sense, this paper presents findings that might be related with possible therapeutic approaches in subsequent studies.

DETAILED DESCRIPTION:
The purpose of the present work was to assess neuromotor abnormalities in aging shoulder. Twenty young adults (20-42), 20 middle-aged adults (43-67) and 20older adults (>68) were recruited. A comparative electromyography (EMG) study was performed on the upper and lower trapezius, middle deltoid, infraspinatus and serratus anterior. The EMG measurement (root mean square (RMS)) and onset time of isometric contractions were analyzed. Body mass index and strength were also tested.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no previously manifested symptoms in the shoulder joint and/or the neck during the past year,

Exclusion Criteria:

* moderate or severe cognitive impairment, rheumatologic diseases, massive osteoarthritis, tumors, shoulder joint instability, circulatory disorders (hemophilia clotting problems) and dermatological problems exacerbated by contact with skin

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants came from Madrid and Castilla La Mancha (Spain) and voluntarily attended the Unit of the Research Group "Physical Therapy in Women´s Health Processes" in the Department of Physical Therapy, University of Alcalá, and the Ocaña Senior Center.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The mean Root Mean Square (RMS) value | 30 minutes
  The electromyographic data were captured simultaneously on a PC by using the LabChart® software. Within the time interval from 2 to 4 seconds after contraction initiation a power spectrum analysis was performed together with the determination of RMS values. The mean RMS values were automatically obtained from the software
onset latency | 30 minutes
  Start of contraction on the basis of 15% of RMS

SECONDARY OUTCOMES:
maximal isometric voluntary contraction | 5 minutes
  Using hand-held dynamometer
body mass index | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Maria Tommes Lacomba, PhD, Study Director — University of Alcalá

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lirio Romero C, Torres Lacomba M, Castilla Montoro Y, Prieto Merino D, Pacheco da Costa S, Velasco Marchante MJ, Bodes Pardo G. Mobilization With Movement for Shoulder Dysfunction in Older Adults: A Pilot Trial. J Chiropr Med. 2015 Dec;14(4):249-58. doi: 10.1016/j.jcm.2015.03.001. Epub 2015 Nov 24. PMID 26793036
- [Result] Phadke V, Camargo P, Ludewig P. Scapular and rotator cuff muscle activity during arm elevation: A review of normal function and alterations with shoulder impingement. Rev Bras Fisioter. 2009 Feb 1;13(1):1-9. doi: 10.1590/S1413-35552009005000012. PMID 20411160
- [Result] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445